CLINICAL TRIAL: NCT00784342
Title: Validation of PROMIS Banks With COPD Exacerbations
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: University of Pittsburgh (Other); Duke University (Other); Endeavor Health (Other)
Responsible Party: Sponsor
Other Study IDs: 07-02
Record Dates: First submitted 2008-10-30; First posted 2008-11-03 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Stable: Patients who are stable have not had a COPD exacerbation in the past 2 months.
- Exacerbation: Patients with an exacerbation have been diagnosed and started on treatment for an exacerbation within the past 3 days.

SUMMARY:
The Patient-Reported Outcomes Measurement Information System (PROMIS) is an NIH Roadmap initiative to develop a computerized system measuring patient-reported outcomes in respondents with a wide range of chronic diseases and demographic characteristics. In the first four years of its existence, the PROMIS network developed item banks for measuring patient-reported outcomes in the areas of pain, fatigue, emotional distress, physical function, and social functioning. During the item banking process, the PROMIS network conducted focus groups, individual cognitive interviews, and lexile (reading level) analyses to refine the meaning, clarity, and literacy demands of all items. The item banks were administered to over 20,000 respondents and calibrated using models based on item response theory (IRT). Using these IRT calibrations, computerized adaptive test (CAT) algorithms were developed and implemented. The network has designed a series of studies using clinical populations to evaluate the item attributes, examine their utility as CATs, and validate the item banks. More information on the PROMIS network can be found at www.nihpromis.org.

DETAILED DESCRIPTION:
This is a prospective longitudinal study of adult patients with chronic obstructive pulmonary disease (COPD) who will be enrolled when their COPD is considered clinically stable or during an acute exacerbation. This design will allow both within-person and between-person comparisons by exacerbation experience. Comprehensive clinical and patient-reported assessments will be performed at baseline and at 3 months (end of study). Subsets of items will be administered by interactive voice response (IVR) over the course of the study to measure changes in key symptoms over the course of recovery from an exacerbation. A subset of patients will be interviewed at the end of the study to assess content validity of PROMIS items in this patient population.

With such a study design, we will be able to evaluate the validity of the PROMIS items in this patient population under acute and stable conditions and evaluate responsiveness of several PROMIS item banks under conditions of known change in an underlying chronic disease. We will also evaluate stability of sub-domains that are not hypothesized to change with COPD exacerbations.

ELIGIBILITY:
Inclusion Criteria:

* An established clinical history of COPD in accordance with the Global Initiative for Chronic Obstructive Lung Disease (GOLD) definition: COPD is a preventable and treatable disease with some significant extrapulmonary effects that may contribute to the severity in individual patients. Its pulmonary component is characterized by airflow limitation that is not fully reversible. The airflow limitation is usually progressive and associated with an abnormal inflammatory response of the lung to noxious particles or gases.
* A history of smoking (at least 10 pack/year history)
* Access to and able to communicate on a touch tone telephone
* Read and speak English
* Able to see and interact with a computer screen, mouse, and keyboard
* A signed and dated written informed consent prior to study participation
* For those enrolled into the exacerbation group: Treatment for an exacerbation may have been started no more than 3 days prior to the day of enrollment for patients recruited in the outpatient setting and no more than 6 days prior to the day of enrollment for patients recruited in the in-patients setting.
* For those enrolled in the stable state group, the patient will be considered stable if he or she has been exacerbation-free for a minimum of 2 months prior to enrollment.

Exclusion Criteria:

* Any concurrent medical or psychiatric condition that may preclude participation in this study or completion of self-administered questionnaires (e.g., moderate to severe dementia and/or severe, uncontrolled schizophrenia, or other condition that would render the participant unable to complete a questionnaire)
* History of asthma without co-existent COPD as the primary diagnosis
* Experiencing a current heart failure exacerbation. (A diagnosis of heart failure is not in itself an exclusion criterion.)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People presenting to primary care or specialty clinics with COPD either with exacerbation or without exacerbation. People admitted to the hospital with a COPD exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren A. Dewalt, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (5):
- United States (5):
  - NorthShore University HealthSystem (Formerly Evanston Northwestern Healthcare), Evanston, Illinois
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Pittsburgh VA Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania